CLINICAL TRIAL: NCT04196894
Title: Ischemic Stroke, Obesity and Thrombolysis (ISOT)
Brief Title: Ischemic Stroke, Obesity and Thrombolysis
Acronym: ISOT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 367/14
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke
Keywords: Thrombolysis; Obesity; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focuses on the relationship between obesity and stroke, which are both characterized by increasing incidence and prevalence with epidemic proportions worldwide and tremendous socio-economic consequences. Furthermore, obesity is an established risk factor for stroke and affects especially younger people, which increases the stroke incidence in younger patients. Unfortunately, the relationship between overweight and acute ischemic stroke including treatment by thrombolysis has not yet been evaluated thoroughly.

DETAILED DESCRIPTION:
All patients receiving thrombolytic treatment for acute ischemic stroke will be included in this study. The decision for treatment and selection of thrombolysis type is allocated to treating stroke physicians who will follow national and international stroke guidelines and considering the clinical and radiological findings. Patients are given either a) intravenous rt-PA (0.9 mg/kg; maximum 90 mg, 10% as intravenous bolus and the remaining 90% as continuous infusion over 1 hour), b) endovascular treatment such as intra-arterial urokinase or rt-PA and/or mechanical recanalization techniques, or c) two thirds of the standard dose intravenous rt-PA followed by endovascular treatment such as intra-arterial urokinase or rt-PA and/or mechanical recanalization techniques (bridging concept). Patient involvement in this study will not influence any treatment decision. Patients will undergo a complete diagnostic stroke work-up, including assessment of vascular risk factors and medication, clinical neurological examination using the National Institutes of Health Stroke Scale (NIHSS) score on admission and 24h after thrombolysis, laboratory examination, brain and neurovascular imaging, echocardiography and 24-hours ECG to determine stroke etiology using the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria. All patients will be weighed as early as possible, but stringently within 24h after thrombolysis. If they are able to stand at 24h, a standard calibrated licensed scale will be used (Seca, Hamburg, Germany; Model 799). Otherwise, patients will be weighed on a special bed scale calibrated and validated for the use for patient weighing (Seca; Hamburg, Germany; Model 657). In addition, body height, waist and hip circumference of each patient will be measured. All patients will be examined by CT and CTA or MRI and MRA at 24h and in any case of clinical deterioration to exclude intracranial hemorrhage and to assess recanalization in case of vessel occlusion (using the thrombolysis in myocardial infarction (TIMI) grading system). The treating physician will initiate secondary prevention of stroke as soon as possible and according to current guidelines. Body weight and clinical assessments (measurement of clinical scores NIHSS, modified Rankin Scale, and Barthel Index; assessment of adverse events such as in-hospital complication, death, cardiovascular event) will be performed by stroke physicians at following visits: I) day 3-5 and/or hospital discharge, II) 3-month and III) 12-month. Patients in whom a clinical follow-up examination is not possible will be evaluated by a structured phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Acute treatment with thrombolysis
* Age >18 years
* Written informed consent

Exclusion Criteria:

* Age <18 years
* Intracranial hemorrhage
* Known hemorrhagic diathesis
* Preexisting neurological deficits (mRS >2 points)
* Uncontrolled arterial hypertension (blood pressure >185/110 mmHg repeatedly despite antihypertensive drugs)
* Severe illness with poor prognosis (e.g. neoplasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving thrombolytic treatment for acute ischemic stroke will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Rates of favourable clinical outcome (mRS 0-2) and death | Month 3

SECONDARY OUTCOMES:
Symptomatic intracranial hemorrhage at 24h after intravenous thrombolysis | Day 1
Recanalisation rates of vessel occlusion at 24h after thrombolysis | Day 1
In-hospital complications | Day 1
Stroke recurrence and myocardial infarction within 12 months after thrombolysis | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Sarikaya, PD Dr.med., Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No